CLINICAL TRIAL: NCT04123288
Title: Single-center, Open-label, Randomized, Two-way Crossover Study to Compare the Single-dose Pharmacokinetics of Pediatric Minitablet and Adult Capsule Formulations of ACT-709478 in Healthy Male Subjects
Brief Title: A Study to Compare a Single-dose of Two Different Formulations of ACT-709478 in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ID-083-104; 2019-002005-22 (EudraCT Number)
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — ACT-709478

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test drug formulation (Experimental): Test drug 60 mg single dose
  Interventions: Drug: ACT-709478
- Reference drug formulation (Active Comparator): 60 mg single dose
  Interventions: Drug: ACT-709478

INTERVENTIONS:
Drug: ACT-709478 — 1 film-coated minitablet contains 2 mg of ACT-709478
  Arms: Test drug formulation
Drug: ACT-709478 — 1 hard capsule contains 10 mg of ACT-709478.
  Arms: Reference drug formulation

SUMMARY:
This study is for research purposes only and is not intended to treat any medical condition. The purpose of this study is to evaluate the pharmacokinetics of 2 different formulations of ACT-709478 in healthy male participants. The participants will be treated in a crossover design with 2 different treatment periods. Pharmacokinetics (PK) is the study of the absorption and breakdown of the study drug in the body.

The duration of participation in this study is approximately 8 weeks from screening to the end of study visit. A screening visit is required within 21 to 3 days prior to the start of the study to determine whether the participant qualifies and is willing to enter in this research study. This study requires the participant to have two in-patient stays in the research clinic. Each in-patient stay is planned for 5 days (4 nights). Eleven days after each dose the participant will have an examination. There will be an in-between period (i.e., time between the end of period 1 and study treatment administration in Period 2) of 7 to 14 days. A safety follow-up telephone call for all participants who have received at least one study treatment will take place 30 to 40 days after the end of study examination or study discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Body mass index of 18.5-28.0 kg/m2 (inclusive) at Screening.
* Czech citizen with the ability to communicate well with the investigator, in a language understandable to the subject, and to understand and comply with the requirements of the study.
* Systolic blood pressure 100 to 145 mmHg, diastolic blood pressure 60 to 90 mmHg, and pulse rate 50 to 90 bpm (inclusive) after 5 min in the supine position at Screening.
* Healthy on the basis of physical examination, cardiovascular assessments, and laboratory tests.

Exclusion Criteria:

* Known hypersensitivity to any of the excipients of the study treatment formulations.
* Participation in a clinical study involving study treatment administration within 3 months or 5 half-lives (whichever is longer) prior to Screening, or in more than 4 clinical studies within 1 year prior to Screening.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatments (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation of the study.
* Any cardiac condition or illness with a potential to increase the cardiac risk of the subject based on medical history, physical examination, or ECG evaluations.
* History or presence of rhythm disorders (e.g., sinoatrial heart block, sick-sinus syndrome, second- or third-degree atrioventricular block, long QT syndrome, symptomatic bradycardia, atrial flutter, or atrial fibrillation).
* PR Interval on 12-lead ECG greater than 200 ms at Screening.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 2 weeks or 5 t½ (whichever is longer) prior to first study treatment administration.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve (AUC 0-t). | Multiple time points; duration for up to 264 hours in each treatment period.
The area under the plasma concentration-time curve (AUC 0-inf) | Multiple time points; duration for up to 264 hours in each treatment period.
The maximum plasma concentration (Cmax) | Multiple time points; duration for up to 264 hours in each treatment period.
The time to reach Cmax (tmax) | Multiple time points; duration for up to 264 hours in each treatment period.
The terminal elimination half-life (t1/2) | Multiple time points; duration for up to 264 hours in each treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- CEPHA s.r.o., Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No